CLINICAL TRIAL: NCT00286832
Title: Evaluation of Response to Treatment Using 18F-FDG Positron Emission Tomography Imaging (PET) With Special Emphasize on the Prognostic Significance of Early On-therapy PET at First-line Treatment in Diffuse Large B-cell Lymphoma Stage IIB-IV
Brief Title: Early On-therapy PET at First-line Treatment in Diffuse Large B-cell Lymphoma Stage IIB-IV
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Nordic Lymphoma Group (Network)
Responsible Party: Lars M Pedersen, MD, Nordic Lymphoma Group (NLG)
Other Study IDs: NLG PET Study
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Diffuse Large-Cell Lymphoma
Keywords: Non-Hodgkin's lymphoma; Diffuse large B-cell lymphoma; PET; Prognosis
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single group study
  Interventions: Procedure: PET scan

INTERVENTIONS:
Procedure: PET scan — One extra PET scan after 1 cycle of treatment.
  Other Names: positron emission tomography

SUMMARY:
Early identification of refractory lymphoma patients provides a basis for stratification between responders to standard approaches and non-responders who may benefit from an early change to an alternative treatment strategy.Metabolic or molecular imaging with fluorine-18 fluorodeoxyglucose positron emission tomography (18F-FDG-PET) has emerged as a powerful imaging modality for diagnosis, staging, and therapy monitoring of a variety of cancers. The primary hypothesis of the present study is that early response can be pinpointed by PET reflecting both tumor burden and activity, as a surrogate for final outcome. An increasing number of studies have suggested the potential role of 18F-FDG PET in the staging and monitoring of lymphomas. The optimal timing of PET scans and the potential role of quantitative PET using SUV to assess response to chemotherapy remain to be defined. Confirmation of very early 18F-FDG-PET as a significant predictor of treatment response in a homogenous group of aggressive lymphoma patients would potentially change the prognosis of the patient by allowing earlier use of alternative therapies and discontinuation of therapy that will not lead to a significant tumour response.

DETAILED DESCRIPTION:
Title: Evaluation of response to treatment using 18F-FDG positron emission tomography imaging (PET) in diffuse large B-cell lymphoma stage IIB-IV with special emphasize on the prognostic significance of early on-therapy PET at first-line treatment

Study design: Multicenter trial.

Planned sample size: 100 patients.

Number of centers: Denmark 2; Sweden 1; Norway 1; Finland 1.

Aim of the study: 1. To evaluate the prognostic significance of PET early after treatment initiation. 2. To compare early PET with standard response criteria for NHL and the International Prognostic Index (IPI) in the prediction of response and outcome.

Primary objective: The prognostic significance of FDG-PET after 1 cycle of chemotherapy.

End-points: Progression-free survival (PFS). Overall survival (OS). Response to treatment (standardized response criteria) at mid-treatment and post-treatment.

Inclusion criteria:

Age ≥ 18 years. Newly diagnosed consecutive patients with diffuse large B-cell lymphoma (DLBCL) according to the WHO classification.

Ann Arbor stage IIB-IV. Written informed consent.

Exclusion criteria: Previously treated with chemotherapy or irradiation. Previous malignant diagnosis except basal cell carcinoma and cervical carcinoma in situ.

Pregnancy. Lactation. Diabetes mellitus. Extreme adipositas. Claustrophobia. Active inflammatory disease or infection.

PET-CT evaluation: PET and CT at primary staging before initiation of therapy and PET after one cycle of intravenous chemotherapy (day 10-20) are mandatory. The results of the PET scans are blinded and will not be available for the local physicians. If the PET result is opened, the patient will be excluded from the study.

Only post-treatment PET scans are allowed outside the protocol. The local physician may use post-treatment PET in diagnostic or therapeutic considerations.

Only dedicated full-ring PET scanners are allowed in this study.

Treatment: Therapy with a CHOP-like backbone according to local standards of the individual centers. Treatment according to other protocols allowed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Newly diagnosed consecutive patients with diffuse large B-cell lymphoma (DLBCL) according to the WHO classification.
* Ann Arbor stage IIB-IV.
* Written informed consent.

Exclusion Criteria:

* Previously treated with chemotherapy or irradiation.
* Previous malignant diagnosis except basal cell carcinoma and cervical carcinoma in situ.
* Pregnancy.
* Lactation.
* Diabetes mellitus.
* Extreme adipositas.
* Claustrophobia.
* Active inflammatory disease or infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample according to the area covered by the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2005-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars M Pedersen, MD, Principal Investigator — Nordic Lymphoma Group (Large Cell Group)
Locations (1):
- Department of Hematology, Odense University Hospital, Odense, Denmark